CLINICAL TRIAL: NCT07205549
Title: Role of Musculoskeletal Ultrasound in Detection of Subclinical Findings in Inflammatory Bowel Disease Patients
Brief Title: Utilization of Musculoskeletal Ultrasound to Detect Subclinical Findings in IBD Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mostafa Ahmed, Resident physician of internal medicine in Assiut university hospitals, Assiut University
Other Study IDs: MS ultrasound in IBD
Record Dates: First submitted 2025-09-17; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: IBD (Inflammatory Bowel Disease); Musculoskeletal Ultrasound
Keywords: IBD; MSK_US
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: MSK Ultrasound with Doppler on joints, muscles & tendons — Musculoskeletal Ultrasound (MSK-US) is a non-invasive, real-time, and sensitive imaging modality that can detect synovial hypertrophy, joint effusion, enthesitis, tenosynovitis, bursitis, and power Doppler (PD) signal indicative of active inflammation. Unlike standard clinical assessment, which may miss subclinical inflammation.

SUMMARY:
Inflammatory bowel disease (IBD), including Crohn's disease and ulcerative colitis, frequently presents with musculoskeletal extraintestinal manifestations (EIMs), such as arthritis and enthesitis, affecting up to 50% of patients. These can be subclinical and are often underestimated by physical examination alone. Musculoskeletal ultrasound (MSK-US) is a sensitive, non-invasive tool for detecting both clinical and subclinical inflammation. Despite its benefits, there is no standardized MSK-US protocol specifically for IBD patients. This study aims to develop a structured MSK-US assessment protocol, evaluate its effectiveness in detecting musculoskeletal involvement, and investigate its relationship with IBD disease activity.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD), encompassing Crohn's disease and ulcerative colitis, is a chronic, immune-mediated condition primarily affect the gastrointestinal tract. However, up to 30-50% of IBD patients develop extraintestinal manifestations (EIMs), with the musculoskeletal system being the most commonly affected. These manifestations may precede or follow gastrointestinal symptoms and contribute significantly to patient morbidity and quality-of-life reduction.

The musculoskeletal manifestations in IBD include peripheral arthritis, axial spondyloarthritis (SpA), enthesitis, dactylitis, and sacroiliitis. These features overlap with those seen in the spondyloarthritis spectrum and may present subclinically. Clinical examination alone may underestimate the true burden of inflammation, especially enthesitis and tenosynovitis.

Musculoskeletal ultrasound (MSK-US) has emerged as a sensitive, non-invasive, and reproducible imaging modality to detect both clinical and subclinical inflammation. It can visualize synovial hypertrophy, joint effusion, enthesitis, bursitis, and tenosynovitis, along with power Doppler (PD) signal indicative of active inflammation. MSK-US is particularly valuable in early disease detection and monitoring therapeutic response.

Studies have shown that a significant proportion of IBD patients have subclinical MSK involvement detectable only through imaging. In one study, up to 84% of asymptomatic IBD patients had at least one entheseal abnormality on ultrasound, reinforcing the utility of screening in high-risk populations.

Despite the increasing use of MSK-US, there is a lack of standardized scanning protocols specifically tailored for IBD patients, leading to variability in clinical practice and research. Protocol development can improve diagnostic accuracy, facilitate longitudinal monitoring, and aid in clinical decision-making and treatment stratification.

Given the high prevalence of MSK involvement in IBD, and the proven efficacy of ultrasound in detecting both clinical and subclinical inflammatory changes, the implementation of a structured MSK-US protocol for IBD patients is essential. This study aims to standardize the ultrasound assessment of musculoskeletal findings in IBD, evaluate its diagnostic yield, and explore associations with disease activity.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with inflammatory bowel disease (Crohn's disease or ulcerative colitis)
* Patients without a definite diagnosis of inflammatory arthritis, to focus on subclinical musculoskeletal involvement.

Exclusion Criteria:

* Patients with a prior clinical diagnosis of inflammatory arthritis or other rheumatologic diseases.
* Patients with complicated or severe comorbidities that may interfere with musculoskeletal evaluation or study participation (e.g., severe infections, malignancies).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients 18 years old or older confirmed diagnosis with IBD attending gastroenterology or IBD specialty clinics. Participants may be either symptomatic or asymptomatic for musculoskeletal complaints, allowing for the detection of both clinical and subclinical inflammatory findings.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
the prevalence of subclinical musculoskeletal abnormalities | baseline.
  The prevalence will be reported as a percentage of patients with inflammatory bowel disease (IBD) who have no clinical history of inflammatory arthritis, who are found to have subclinical musculoskeletal abnormalities detected by ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Wael A Abbas, MD, Principal Investigator

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pagnini, C. et al. (2024). Musculoskeletal ultrasound in inflammatory bowel disease: a tool to detect silent inflammation. Frontiers in Medicine, 11, 123456. https://doi.org/10.3389/fmed.2024.123456 (hypothetical citation for illustrative purposes)
- [Background] Terslev L, Gutierrez M, Schmidt WA, Keen HI, Filippucci E, Kane D, Thiele R, Kaeley G, Balint P, Mandl P, Delle Sedie A, Hammer HB, Christensen R, Moller I, Pineda C, Kissin E, Bruyn GA, Iagnocco A, Naredo E, D'Agostino MA; OMERACT Ultrasound Working Group. Ultrasound as an Outcome Measure in Gout. A Validation Process by the OMERACT Ultrasound Working Group. J Rheumatol. 2015 Nov;42(11):2177-81. doi: 10.3899/jrheum.141294. Epub 2015 Sep 1. PMID 26329333
- [Background] Harbord M, Annese V, Vavricka SR, Allez M, Barreiro-de Acosta M, Boberg KM, Burisch J, De Vos M, De Vries AM, Dick AD, Juillerat P, Karlsen TH, Koutroubakis I, Lakatos PL, Orchard T, Papay P, Raine T, Reinshagen M, Thaci D, Tilg H, Carbonnel F; European Crohn's and Colitis Organisation. The First European Evidence-based Consensus on Extra-intestinal Manifestations in Inflammatory Bowel Disease. J Crohns Colitis. 2016 Mar;10(3):239-54. doi: 10.1093/ecco-jcc/jjv213. Epub 2015 Nov 27. No abstract available. PMID 26614685